CLINICAL TRIAL: NCT05987345
Title: Safety and Clinical Efficacy Evaluation of Pulsed Electric Field Therapy in Patients With Late-stage Non-small Cell Lung Cancer
Brief Title: Trial of Pulsed Electric Field Therapy in Patients With Late-stage Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Energenx Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCFIM-001
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: NSCLC
Keywords: NSCLC; PEF; Immune Checkpoint Inhibitor(ICI)
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEF treatment (Experimental): All of participants who signed the Informed Consent Form(ICF) and meet all of inclusion and exclusion criterial will be enrolled to experimental arm. PEF treatment on Day 1, followed by anti PD-1 on Day 7 and then routinely.
  Interventions: Device: PEF; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Device: PEF — PEF device treated in the trial.
Drug: Anti-PD-1 monoclonal antibody — Anti-PD-1 monoclonal antibody administered on Day 7 then routinely.

SUMMARY:
The goal of this clinical trial is to verify the safety and clinical benefit of pulsed electric field(PEF) treatment of metastatic non-small cell lung cancer(NSCLC) patients with acquired resistance to anti programmed cell death protein 1(PD-1) monoclonal antibody therapy.

The main questions it aims to answer are:

* Safety of PEF treatment of metastatic NSCLC patients.
* Control of ablated and other targeted lesions.
* Local and peripheral immunoregulation effect. PEF energy will be delivered to preselected lesions of participants, then anti PD-1 will be routinely administrated if no adverse event(AE)/serious adverse event(SAE) which need medical intervention occurs.

DETAILED DESCRIPTION:
Eligible patients will will be enrolled to experimental arm and receive standard of care combining with PEF treatment on Day 1, followed by anti PD-1 on Day 7 and then routinely.

All kinds of adverse events will be recorded and analyzed to evaluate the safety of the treatment. At the same time, the local control rate of treated lesions, PFS and OS after PEF will be analyzed to evaluate the clinical value of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 22 years old with pathologically confirmed non-small cell lung cancer stage III-IV.
2. Patients received first-line anti PD-1 immunotherapy and had disease progression.
3. Lesions to be ablated must be ≤ 3cm in longest diameter(LD).

   * The leison to be ablated can be ≤ 5cm in LD, if evaluated as possible with multiple energy delivery in a single session.
4. More than one measurable lesion according to RECIST 1.1 except PEF targeted lesions.
5. Eastern Cooperative Oncology Group(ECOG) performance status 0-1
6. Life expectancy ≥3 months
7. Fully understand the treatment plan and sign the informed consent form voluntarily.

Exclusion Criteria:

1. Patients should be excluded if they received surgery within 30 days.
2. Patients should be excluded if they received any form of local treatment within 30 days.
3. Accompanied by uncontrolled metastasis of the central nervous system.
4. Have a history of severe adverse reactions to ICI.
5. With uncontrolled immune system diseases or being treated with immunosuppressants.
6. Severe abnormality of liver and kidney function, which was evaluated by the researchers as unsuitable for admission.
7. Patients with abnormal blood coagulation and antiplatelet therapy due to cardiovascular and cerebrovascular diseases should be discontinued one week before PEF treatment according to the evaluation of clinicians.
8. Accompanied by infectious diseases that cannot be effectively controlled.
9. Suffered from other severe lung diseases (including interstitial pneumonia, pulmonary fibrosis, pulmonary fibrosis with emphysema, atelectasis, etc.)
10. Patients who had severe cardiac dysfunction and had a history of arrhythmias in the past 2 years, including rapid atrial arrhythmias, any rapid ventricular arrhythmias, a history of degree II or III atrioventricular block, and sinus bradycardia with a heart rate of less than 45 beats per minute.
11. Patients who are participating in other clinical trials.
12. With a cardiac pacemaker or metal implant in the chest.
13. Women who are pregnant or lactating, or who plan to become pregnant during the study.
14. The researchers determined that there were other conditions in which patients were not suitable for enrollment.
15. Patients who have a history of receiving non-first-line anti PD-1 immunotherapy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Technical success rate of PEF treatment | 7 days
  The percentage of the number that the equipment successfully reached the target lesion and completed PEF energy delivery.
Incidence of PEF treatment related AE/SAEs | 1 month
  The incidence and severity of PEF treatment related adverse events according to CTCAE version 4.0

SECONDARY OUTCOMES:
Local control of ablated lesions by CT | 3 months
  Compared with the baseline CT scan before treatment, the maximum diameter of the ablated lesion decreased, remained unchanged or increased by less than 20%.
Local control of ablated lesions by CT | 6 months
  Compared with the baseline CT scan before treatment, the maximum diameter of the ablated lesion decreased, remained unchanged or increased by less than 20%.
Progression free survival rate at 6 months | 6 months
Overall survival rate at 6 months | 6 months
Overall survival rate at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, MD, Principal Investigator — The first Affiliated Hospital of Guanzhou Medical University
Locations (1):
- The first Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China